CLINICAL TRIAL: NCT05344053
Title: Development and Assessment of the Precise Management and Rehabilitation Model of Coronary Artery Disease Under the Hierarchical Medical System
Brief Title: Community-based Precise Management for Patients With Coronary Artery Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Haiyan Xu, Chief Physician, MD, PhD, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: XCSTS-SD2020-11
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Risk Factor Control; Community-based Management; Secondary Prevention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community-based precise management (Experimental)
  Interventions: Other: Community-based precise management
- Standard community-based management (Active Comparator)
  Interventions: Other: Standard community-based management

INTERVENTIONS:
Other: Community-based precise management — The community-based precise management is a modified management strategy beyond the traditional standard community-based care under the hierarchical medical system of China. In the intervention arm, the community doctors receive training to improve their skills on coronary artery disease management. Patients will be under management for 1 year according to the strategies of community-based precise management and rehabilitation model.
  Arms: Community-based precise management
Other: Standard community-based management — The standard community-based management is the usual community-based care under the hierarchical medical system of China. In this arm, the community doctors will not receive any training on precise management strategies to improve their skills on coronary artery disease management, and patients will be under usual care for 1 year.
  Arms: Standard community-based management

SUMMARY:
The community-based precise management for patients with coronary artery disease study is a prospective, cluster-randomized, open-labeled trial. The purpose of this trial is to test whether a community-based precise management and rehabilitation model under the hierarchical medical system could help improve the cardiovascular risk factors control in patients with coronary artery disease. Additionally, the trial will also evaluate the impact of the model on major cardiovascular adverse events in patients with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with prior myocardial infarction
* or receiving percutaneous coronary intervention or coronary artery bypass graft;
* or coronary artery stenosis≥50% defined by coronary angiography or coronary CT angiography

Exclusion Criteria:

* Refuse to sign the written informed consent;
* Patients without the ability to take care of themselves;
* Mental disorders;
* Alcoholics or drug addicts;
* Cannot be followed up for any reasons;
* Life expectancy<1 year due to non-cardiovascular reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Status of risk factors control of coronary artery disease | 1 year
  A composite of not smoking, blood pressure<140/90mmHg/<130/80mmHg for patients with diabetes, HbA1c≤7%, LDL-C<1.8mmol/L, antiplatelet therapy, and statins use.

SECONDARY OUTCOMES:
All-cause death | 1 year
Readmission | 1 year
Myocardial infarction | 1 year
Coronary revascularization | 1 year
Stroke | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Infirmary of Industrial and Commercial Bank of China, Beijing, Beijing Municipality, China